CLINICAL TRIAL: NCT04332120
Title: Comparison of Results of Different Surgical Techniques Used in Female Tubal Sterilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alanya Alaaddin Keykubat University (Other)
Responsible Party: Principal Investigator, muhammet serhat yıldız, Gynecologist and Obstetrician, Principal Investigator, Alanya Alaaddin Keykubat University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 82752631
Record Dates: First submitted 2020-03-30; First posted 2020-04-02 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Sterilization, Tubal; Visual Analog Pain Scale
Keywords: colpotomy; sterilization; VAS; contraception
MeSH Terms: interventions — Sterilization, Tubal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mini Laparotomic (Active Comparator): In patients undergoing spinal anesthesia, a suprapubic 3-5 centimeter incision was entered into the abdomen. After both tubes were isolated, bilateral tube ligation was performed by Pomeroy method. After bleeding control was achieved, it was repaired in accordance with the anatomy of the abdomen.
  Interventions: Procedure: tubal sterilization
- Laparoscopic (Active Comparator): In patients undergoing general anesthesia, Verres was inserted into the abdomen through the umbilicus. Pneumo peritoneum was created with carbon dioxide (CO2). Optical imaging was placed into the abdomen from the umbilicus with 10-trochar. Auxiliary trochars from 3 centimeter supero-medial of both spina iliaca anterior superior were placed in the abdomen. bilateral tubas were isolated. Bilateral tubal ligation was performed with the help of bipolar cautery. bleeding control was achieved. trochars were taken out of the abdomen. the skin was closed.
  Interventions: Procedure: tubal sterilization
- posterior colpotomy (Active Comparator): The patient underwent spinal anesthesia and was placed in a high lithotomy position. cervical uteri was observed with the help of speculum. A 3 centimeter vertical incision was opened 2 centimeter below the cervix uteri. Peritoneal cavity was entered from this area. bilateral tubas were isolated. Bilateral tubal ligation was performed using the pomeroy method. bleeding control was achieved. peritoneal and posterior cervical incision line was repaired.
  Interventions: Procedure: tubal sterilization

INTERVENTIONS:
Procedure: tubal sterilization

SUMMARY:
The investigator's aim in this study is to compare the results of tubal ligation surgery, one of the contraceptive methods, between different surgical techniques. 194 patients were included in the study. Of these patients, 104 had vaginal approach, 44 had laparotomic and 46 had laparoscopic tube ligation surgery. These surgical techniques are statistically was compared; Visual Analog Pain Scale (VAS) after surgery, in terms of duration of surgery, length of hospital stay, cost to hospital and amount of blood loss. As a result of the analysis; tubal sterilization technique performed with vaginal colpotomy were found to be more successful than other techniques; Visual Analog Pain Scale score, postoperative hospital stay, operation time and cost.

DETAILED DESCRIPTION:
The study compared the peroperative effects and postoperative results of different surgical techniques with three different techniques in patients undergoing tubal sterilization.

surgical techniques used:

1. Mini Laparotomic tubal ligation
2. Laparoscopic tubal ligation
3. tubal ligation by posterior colpotomy

A total of 194 patients were included in the study. Tubal ligation was performed in 44 patients with mini laparotomy, 46 patients with laparoscopy and 104 patients with posterior colpotomy technique.

The following parameters were evaluated in the study

1. Parity
2. How many of their previous births are vaginal delivery, how many are cesarian section
3. 6th hour Visual Analog Pain Scale (VAS) score
4. 24th hour Visual Analog Pain Scale (VAS) score
5. Preoperative - postoperative hmg differences
6. Surgery time
7. Length of hospital stay

ELIGIBILITY:
Inclusion Criteria:

* Over 31 years old
* Have completed the fertility request
* Accepting informed consent

Exclusion Criteria:

* Being under the age of 32
* Having a child desire

Min Age: 32 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — an operation for female
Enrollment: 194 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Pain Scale (VAS) | postoperative 6th hour
  postoperative pain degree. 0-10 point. 0 worst, 10 best
Visual Analog Pain Scale (VAS) | postoperative 24th hour
  postoperative pain degree. 0-10 point. 0 worst, 10 best
the amount of bleeding | 24 hour
  preoperative and postoperative hemogram differences
length of hospital stay | 48 hour
  postoperative hospitalization
duration of surgery | minimum duration of surgery 15 minute, maximum duration of surgery 60 minute
  The time from the administration of anesthesia to the end of the operation

CONTACTS AND LOCATIONS:
Overall Officials: serhat yıldız, Study Director — AKU

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] American College of Obstetricians and Gynecologists' Committee on Practice Bulletins-Gynecology. ACOG Practice Bulletin No. 208: Benefits and Risks of Sterilization. Obstet Gynecol. 2019 Mar;133(3):e194-e207. doi: 10.1097/AOG.0000000000003111. PMID 30640233
- [Background] Schlaeder G, Boudier E. [Tubal sterilization]. Rev Prat. 2002 Oct 15;52(16):1790-4. French. PMID 12564171
- [Background] Chang WH, Liu JY, Yeh YC, Wu GJ, Chiang YJ, Yu MH, Chen CH. Tubal ligation via colpotomy or laparoscopy: a retrospective comparative study. Arch Gynecol Obstet. 2011 Apr;283(4):805-8. doi: 10.1007/s00404-010-1435-z. Epub 2010 Mar 26. PMID 20339859
- [Background] Harkki-Siren P, Sjoberg J, Kurki T. Major complications of laparoscopy: a follow-up Finnish study. Obstet Gynecol. 1999 Jul;94(1):94-8. PMID 10389725